CLINICAL TRIAL: NCT02664012
Title: A Single-Center, Randomized, Open-Label, Crossover Study to Assess Elements of Abuse Liability for Three Menthol Electronic Cigarettes
Brief Title: Comparison of Nicotine Plasma Concentrations and Subjective Effects for Three Menthol Electronic Cigarettes vs Combustible Menthol Cigarettes and Nicotine Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R.J. Reynolds Vapor Company (Industry)
Collaborators: Celerion (Industry); RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD1501
Record Dates: First submitted 2016-01-13; First posted 2016-01-26 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Smoking
Keywords: adoption; electronic cigarettes; e-cigarettes; menthol; combustible cigarettes; nicotine polacrilex; own brand cigarette; subjective measures; pharmacokinetics; pharmacodynamics; cigarette
MeSH Terms: conditions — Smoking; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Own Brand Menthol Cigarette (Active Comparator): Own Brand Menthol Cigarette
  Interventions: Other: Own Brand Menthol Cigarette
- Electronic Menthol Cigarette #1 (Experimental): VUSE® (menthol flavor, 14 mg nicotine)
  Interventions: Other: Electronic Menthol Cigarette #1
- Electronic Menthol Cigarette #2 (Experimental): VUSE® (menthol flavor, 29 mg nicotine)
  Interventions: Other: Electronic Menthol Cigarette #2
- Electronic Menthol Cigarette #3 (Experimental): VUSE® (menthol flavor, 36 mg nicotine)
  Interventions: Other: Electronic Menthol Cigarette #3
- Leading U.S. Nicotine Gum (Active Comparator): 4 mg nicotine polacrilex gum
  Interventions: Other: Leading U.S. Nicotine Gum

INTERVENTIONS:
Other: Own Brand Menthol Cigarette — combustible menthol cigarette brand style smoked most frequently by subject
  Arms: Own Brand Menthol Cigarette
Other: Electronic Menthol Cigarette #1 — VUSE® Digital Vapor Cigarette (menthol flavor, 14 mg nicotine)
  Arms: Electronic Menthol Cigarette #1
Other: Electronic Menthol Cigarette #2 — VUSE® Digital Vapor Cigarette (menthol flavor, 29 mg nicotine)
  Arms: Electronic Menthol Cigarette #2
Other: Electronic Menthol Cigarette #3 — VUSE® Digital Vapor Cigarette (menthol flavor, 36 mg nicotine)
  Arms: Electronic Menthol Cigarette #3
Other: Leading U.S. Nicotine Gum — 4 mg nicotine polacrilex gum
  Arms: Leading U.S. Nicotine Gum

SUMMARY:
The purpose of this study is to measure plasma nicotine uptake parameters, physiological measures, and subjective effect measures in smokers during and following a single ad libitum use of three menthol electronic cigarettes versus combustible menthol cigarettes and nicotine gum.

DETAILED DESCRIPTION:
This study will assess various elements that may provide information regarding the potential for menthol electronic cigarettes (e-cigarettes) to be adopted by current smokers. These various elements include: a) nicotine pharmacokinetics (PK), b) physiological measures of pulse rate and blood pressure, and c) subjective effects measured by Urge to Smoke, Urge for Product, Product Rating, Intent to Use Product Again, and Product Effects.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form and complete questionnaires written in English.
2. Generally healthy male or female, 21 to 60 years of age, inclusive, at Screening.
3. Expired breath carbon monoxide (ECO) level is ≥ 15 ppm and ≤ 100 ppm at the Screening and Randomization Visits, measured between 12 p.m. and 6 p.m.
4. Combustible menthol cigarettes are the only tobacco product used within (≤) 30 days of Screening.
5. Smokes combustible, filtered, menthol cigarettes, 83 mm to 100 mm in length.
6. Agrees to smoke usual brand (UB) menthol cigarette throughout the study period. Usual brand cigarette is defined as the menthol cigarette brand style currently smoked most frequently by the subject.
7. Smokes at least 10 menthol cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the Investigator.
8. Response at Screening to Fagerstrom Test for Nicotine Dependence, Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6 - 30 minutes."
9. Willing to use UB menthol cigarette, the study electronic cigarette menthol brand styles and nicotine gum during the study period.
10. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to check-in at each Test Visit.
11. Females of childbearing potential must be willing to use a form of contraception acceptable to the Investigator from the time of signing informed consent until study discharge.

Exclusion Criteria:

1. Clinically significant or unstable/uncontrolled acute or chronic medical conditions at Screening, as determined by the Investigator, that would preclude a subject from participating safely in the study (e.g., uncontrolled hypertension, asthma or other lung disease, cardiac disease, neurological disease or psychiatric disorders) based on safety assessments such as clinical laboratory tests, medical history, and physical/oral examinations.
2. Systolic blood pressure of > 150 mmHg or a diastolic blood pressure of > 95 mmHg at Screening, measured after being seated for at least 5 minutes.
3. Hemoglobin level is < 12 g/dL at Screening.
4. Positive test for Human Immunodeficiency Virus (HIV), Hepatitis B surface antigen, or Hepatitis C virus.
5. Postponing a decision to quit smoking (defined as planning a quit attempt within [≤] 30 days of Screening) to participate in this study or previous attempt within (≤) 30 days prior to Screening.
6. Employed by a tobacco company, the study site, or handles unprocessed tobacco as part of their job.
7. Use of any medication or supplement that aids smoking cessation, including but not limited to any nicotine replacement therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix), bupropion (Wellbutrin, Zyban), or lobelia extract within (≤) 30 days of Screening.
8. Females ≥ 35 years of age currently using systemic, estrogen containing contraception or hormone replacement therapy.
9. A positive urine drug screen without disclosure of corresponding prescribed concomitant medication(s), at Screening or Randomization Visit. A positive alcohol result at Screening, Randomization Visit, or at any Test Visit.
10. A female who is pregnant, lactating, or intends to become pregnant during the course of the study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Nicotine pharmacokinetics with respect to initiation of in-clinic investigational product (IP) use following a 12-hour tobacco and nicotine abstinence | -5, -0.5, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300, 360 minutes
  Determine area under the plasma nicotine concentration versus time curve (AUC)
Nicotine pharmacokinetics with respect to initiation of in-clinic investigational product (IP) use following a 12-hour tobacco and nicotine abstinence | -5, -0.5, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300, 360 minutes
  Determine maximum plasma nicotine concentration (Cmax), baseline adjusted
Nicotine pharmacokinetics with respect to initiation of in-clinic investigational product (IP) use following a 12-hour tobacco and nicotine abstinence | -5, -0.5, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300, 360 minutes
  Determine time to maximum plasma nicotine concentration (Tmax), baseline-adjusted
Subjective effects scores for Urge to Smoke (UTS) with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | -10, 5, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360 minutes
  Score subjective effects using a numeric rating scale (NRS) to determine area under the UTS score-versus-time curve [area under the effect curve (AUEC)]
Subjective effects scores for Intent to Use Again (IUA) with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | 15, 30, 45, 60, 120, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine area under the IUA score-versus-time curve (AUEC)
Subjective effects scores for Product Ratings (PR) with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | 15, 30, 45, 60, 120, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine area under the PR score-versus-time curve (AUEC)
Subjective effects scores for Positive Product Effects (PE) with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | 15, 30, 45, 60, 120, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine area under the Positive PE score-versus-time curve (AUEC)
Subjective effects scores for Negative Product Effects (PE) with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | 15, 30, 45, 60, 120, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine area under the Negative PE score-versus-time curve (AUEC)
Maximum change in pulse rate relative to baseline | Baseline and at timed intervals over 360 minutes following initiation of IP use
  Determine the maximum change in pulse rate
Baseline cotinine measured pre-IP use | -0.5 minute (baseline) and -5 min (back-up baseline) for each IP
  Evaluate changes in baseline cotinine to assess whether subjects substantially changed their nicotine uptake during the study
Change in expired carbon monoxide (ECO) relative to baseline | Baseline and 35 minutes post-IP use
  Assess change in ECO from baseline following IP use
Subjective effects scores for UTS with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | -10, 5, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine minimum UTS score
Subjective effects scores for UTS with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | -10, 5, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine time to minimum UTS score
Subjective effects scores for IUA with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | 15, 30, 45, 60, 120, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine maximum IUA score
Subjective effects scores for PR with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | 15, 30, 45, 60, 120, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine maximum PR score
Subjective effects scores for Positive PE with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | 15, 30, 45, 60, 120, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine maximum Positive PE score
Subjective effects scores for Negative PE with respect to initiation of in-clinic IP use following a 12-hour tobacco and nicotine abstinence | 15, 30, 45, 60, 120, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine maximum Negative PE score

OTHER OUTCOMES:
Maximum change in blood pressure relative to baseline | Baseline and at timed intervals over 360 minutes following initiation of IP use
  Determine the maximum change in blood pressure
Subjective effects scores for Urge for Product (UFP) with respect to initiation of in-clinic IP use (e-cigarettes and nicotine gum only) following a 12-hour tobacco and nicotine abstinence | -10, 5, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine area under the UFP score-versus-time curve (AUEC)
Subjective effects scores for UFP with respect to initiation of in-clinic IP use (e-cigarettes and nicotine gum only) following a 12-hour tobacco and nicotine abstinence | -10, 5, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine maximum UFP score
Subjective effects scores for UFP with respect to initiation of in-clinic IP use (e-cigarettes and nicotine gum only) following a 12-hour tobacco and nicotine abstinence | -10, 5, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360 minutes
  Score subjective effects using a NRS to determine time to maximum UFP score
Perform CYP2A6 genotyping | Once, at time of randomization
  A) Assess the impact of CYP2A6 genotype on nicotine uptake and subjective effects following a 12-hour tobacco and nicotine abstinence and B) Explore a potential relationship between CYP2A6 genotype and phenotype
Perform phenotyping (i.e., nicotine metabolic ratio of cotinine:3-hydroxy cotinine) | Once, at time of randomization
  A) Assess the impact of phenotypic ratio on nicotine uptake and subjective effects following a 12-hour tobacco and nicotine abstinence and B) Explore a potential relationship between CYP2A6 genotype and phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gartner, MD, Principal Investigator — Celerion; Charles Tomek, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stiles MF, Campbell LR, Jin T, Graff DW, Fant RV, Henningfield JE. Assessment of the abuse liability of three menthol Vuse Solo electronic cigarettes relative to combustible cigarettes and nicotine gum. Psychopharmacology (Berl). 2018 Jul;235(7):2077-2086. doi: 10.1007/s00213-018-4904-x. Epub 2018 May 3. PMID 29725702